CLINICAL TRIAL: NCT06330701
Title: Post-Operative Outcomes Following the Treatment of Kidney Stones With the MONARCH Platform, Urology
Brief Title: Stone Access and Removal (STAR) Study
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023URO0001; 2023URO0001 (Other: Auris Health,Inc.)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Kidney Calculi
Keywords: Nephrolithotomy; Percutaneous; Ureteroscopy; Robotic; Monarch; Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic mini-Percutaneous Nephrolithotomy (PCNL) (Experimental): Participants with kidney stones will be enrolled for a robotic-assisted mini-percutaneous nephrolithotomy procedure using the MONARCH Platform, Urology for removal of kidney stones. The MONARCH Platform, Urology enables electro-mechanical articulation and precise control of a flexible ureteroscope and/or a flexible mini-PCNL suction catheter ("catheter") for visualization and access to the urinary tract for diagnostic and therapeutic procedures.
  Interventions: Device: Robotic-assisted mini-PCNL

INTERVENTIONS:
Device: Robotic-assisted mini-PCNL — This robotically enabled hybrid procedure called the MONARCH Mini-PCNL will allow the clinician to obtain retrograde and percutaneous access to participant's kidney under continuous visualization for therapeutic applications (i.e., stone removal).

SUMMARY:
The purpose of the study is to assess procedural completion, the post-operative stone clearance and the safety profile following robotic mini-Percutaneous Nephrolithotomy (PCNL) performed with the MONARCH Platform, Urology.

ELIGIBILITY:
Inclusion Criteria:

* Simple renal caliceal and/or pyelo stone(s) with stone burden => 1 cm, identified on CT scan, and appropriate for PCNL treatment according to AUA guidelines
* Normal upper tract anatomy, amenable to PCNL and ureteroscopy
* Participants with a percutaneous tract length < 15 cm as measured by the estimation of the skin to stone or skin to appropriate calyx for treatment through a CT scan
* Participant is an appropriate candidate for a mini-PCNL based on the clinical guidelines and investigator assessment.

Exclusion Criteria:

Pre-Procedure:Exclusion Criteria:

* Any medical or physical condition/limitation that would contra-indicate a conventional ureteroscopy or PCNL in the supine position (e.g., atypical interposition of visceral organs (bowel, spleen, or liver))
* Expected additional procedure, or participation in any clinical trial, from 30 days prior to the study procedure and throughout the duration of the study, which might impact this study's results
* A solitary functioning kidney
* Female participants who are pregnant or nursing or those of child-bearing potential refusing a pregnancy test
* Presence of ureteral impacted stones

Intra-Procedure Exclusion Criteria:

- Any presenting condition discovered intra-procedurally that in the opinion of the investigator would make participating in this study not in the participant's best interest.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Robotic-assisted mini-Percutaneous Nephrolithotomy (PCNL) Kidney Stone Removal Procedure Completed | Procedure Visit (Day 0)
  The percentage of Robotic-assisted mini-PCNL procedures that are successfully completed will be reported. Completion is defined as: (1) gained safe concomitant (that is, retrograde and antegrade) access to the upper urinary tract, (2) located and visualized kidney stones, (3) enabled fragmentation of stones by standard of care method (4) evacuated stone fragments and dust, and (5) Complete treatment without need for case conversion, as assessed by the investigator.

SECONDARY OUTCOMES:
Stone Free Rate (%) | Post-operative Day 30
  Stone free is defined as having <= 4mm residual stones detected by computed tomography (CT), assessed at post-operative Day 30.
Number of Adverse Events | Up to post-operative Day 90
  Adverse events are defined as any undesirable clinical occurrence in a participant, whether or not it is considered to be device-related.
Number of Procedure Conversions to Conventional Treatment Methods due to study device-related safety event | Procedure Visit, Day 0
  Number of procedures converted to conventional stone removal procedures (e.g., ureteroscopy or percutaneous nephrolithotomy) due to the occurrence of a study device-related safety event.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A. Knoedler, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - UW School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No